CLINICAL TRIAL: NCT00227786
Title: Using Electronic Medical Records to Measure and Improve Adherence to Tobacco Treatment Guidelines in Primary Care
Brief Title: Primary Care Physicians' Use of Stop-Smoking Plans to Help Patients Who Are Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CDR0000448865; KAISER-U19-CA099193
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2005-11

CONDITIONS: Tobacco Use Disorder; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; tobacco use disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: smoking cessation intervention
Other: counseling intervention

SUMMARY:
RATIONALE: Stop-smoking plans suggested by physicians may help patients quit smoking. Studying how physicians give stop-smoking treatment as family doctors may increase the chance of smokers receiving such treatment.

PURPOSE: This randomized clinical trial is studying physicians' practice patterns to see if regular feedback to the physician increases the chance of adult smokers receiving stop-smoking treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop an automated coding system using existing electronic medical records (EMRs) to assess adherence to national tobacco-cessation treatment guidelines by individual physicians in the primary care setting at 4 health maintenance organizations.
* Compare the validity of the automated coding system with that of coding performed by medical record abstractors.
* Determine the effect of performance feedback on tobacco treatment practice patterns over 2 years among primary care physicians.
* Provide recommendations for recording tobacco-cessation treatment services in EMR systems and evaluating adherence to treatment guidelines.
* Produce a set of computer programs that can be easily adopted in diverse health care settings for assessing adherence to the national tobacco-cessation treatment guidelines using data from EMRs.

OUTLINE: This is a randomized, controlled, multicenter study. Physicians from each participating center are sorted into pairs according to their rate of providing advice to quit smoking to identified adult smokers and the number of identified adult smokers seen in the 3-month baseline observation period. Each physician in the pair is then randomized to 1 of 2 arms.

* Arm I (automated coding system feedback): Physicians receive reports from an automated coding system regarding their performance in administering tobacco-cessation services in each of the five A's (Ask, Advise, Assess, Assist, and Arrange) to identified smokers in comparison with their past performance and in comparison with their anonymous colleagues once every 3 months. One year after randomization, these physicians are further randomized, using the same paired-group approach, to either continue receiving automated coding system feedback for 1 additional year OR to stop receiving feedback.

Physicians receive a survey at the end of 2-year period regarding the usefulness of each aspect of the feedback reports and the feedback program in general.

* Arm II (control): Physicians do not receive any information regarding their performance in administering tobacco-cessation services in each of the five A's to identified smokers.

A questionnaire about tobacco-cessation services in primary care is sent to patients of all physicians within two weeks of each patient's primary care visit and then at the end of the first year of providing feedback to physicians to compare patient report of tobacco-cessation services with what is documented in the electronic medical record for that primary care visit.

PROJECTED ACCRUAL: At least 40 primary care physicians per participating center and 1,000 patients (250 per participating center) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Primary care physician, meeting all of the following criteria:

  * Practicing medicine in a family practice or internal medicine clinic
  * Scheduled to see adult primary care patients for ≥ 2½ days (or 5 half days or equivalent combination of full and half days) per week
  * Planning to continue full-time practice in their participating organization for at least the next 2 years
  * At least 1 year of experience working with the local electronic medical record system
* Patient

  * Adult smoker who visited a study physician within the past month

PATIENT CHARACTERISTICS:

Age

* Adult

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2003-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change in tobacco cessation care delivery of the 5 A's (Ask, Advise, Assess, Assist, and Arrange) and in the percentage of smokers receiving assistance as measured by MediClass classification at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Victor J. Stevens, PhD, Study Chair — Kaiser Permanente
Locations (5):
- United States (5):
  - Kaiser Permanente - Aurora, Aurora, Colorado
  - Kaiser Permanente Center for Health Research - Hawaii, Honolulu, Hawaii
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Harvard Pilgrim Health Care, Boston, Massachusetts
  - Kaiser Permanente Center for Health Research, Portland, Oregon